CLINICAL TRIAL: NCT00763035
Title: Comparison of Dobutamine and Regadenoson Stress CMR
Brief Title: Comparison of Dobutamine and Regadenoson Stress Cardiac Magnetic Resonance (MR)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Potential participants with COPD/asthma unwilling to participate.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00006484
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease; Asthma; Chronic Obstructive Pulmonary Disease (COPD); Angina
Keywords: Coronary Artery Disease; Coronary Vessels; Myocardial Ischemia; Coronary Disease; Ischemic heart disease; asthma; copd
MeSH Terms: conditions — Coronary Artery Disease; Asthma; Pulmonary Disease, Chronic Obstructive; Angina Pectoris; Myocardial Ischemia; Coronary Disease | interventions — regadenoson; Dobutamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): Arm A will get Dobutamine Stress test with cardiac MR (CMR). Both arms will then cross over to the other arm to get the second test. So each participant will undergo two types of testing.
  Interventions: Drug: Regadenoson; Drug: Dobutamine
- B (Active Comparator): Arm B will get Regadenoson stress test with CMR. Both arms will then cross over to the other arm to get the second test. So each participant will undergo two types of testing.
  Interventions: Drug: Regadenoson; Drug: Dobutamine

INTERVENTIONS:
Drug: Regadenoson — Each participant will receive regadenoson 0.4mg (5ml) one time bolus dose at one visit.
  Other Names: Lexiscan
Drug: Dobutamine — Each participant will receive dobutamine infusion (as per protocol to achieve a target heart rate of 85% of predicted for age) at another visit.
  Other Names: Dobutrex

SUMMARY:
The goal of this research is to determine the utility of Regadenoson (Lexiscan)for use as an imaging agent with cardiac MR. If found useful, it will help us establish a protocol for regadenoson stress MR perfusion (Regadenoson stress test with cardiac MR).The investigators will compare regadenoson with dobutamine so each participant will undergo two studies. A cardiac MR stress test with regadenoson and with dobutamine. The investigators participants will include patients with history of COPD and Asthma, so it will also help us determine feasibility of Regadenoson in these patient's subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40 to 85 years with OBSTRUCTIVE AIRWAY DISEASES (ASTHMA AND COPD) and a forced expiratory volume (FEV1) > 0.5.
* Patients should have a clinical indication to undergo cardiac stress test with dobutamine.

Exclusion Criteria:

* Those with pacemakers, defibrillators, functioning neural stimulator devices or other implanted electronic devices.
* Ferromagnetic cerebral aneurism clips or other intraorbital and intracranial metal.
* An allergy to Gadolinium or other severe drug allergies.
* Acute myocardial infarction within 3 months.
* Moderate or severe aortic stenosis or other significant valvular disease;
* Claustrophobia.
* High grade (2o or 3o) AV Block.
* Closed angle glaucoma.
* Participants unable to provide informed consent.
* Renal dialysis (subjects with moderate-to-severe renal impairment defined as eGFR < 60 mL/min.
* A contraindication to receipt of dobutamine.
* Participants with known coronary artery disease will be included with the exception that patients with left main or narrowings >50% in the distributions of the left anterior descending, circumflex, and right coronary artery will be excluded.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Hundley, M.D., F.A.C.C., F.A.H.A, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- WAKE FOREST UNIVERSITY Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Leaker BR, O'Connor B, Hansel TT, Barnes PJ, Meng L, Mathur VS, Lieu HD. Safety of regadenoson, an adenosine A2A receptor agonist for myocardial perfusion imaging, in mild asthma and moderate asthma patients: a randomized, double-blind, placebo-controlled trial. J Nucl Cardiol. 2008 May-Jun;15(3):329-36. doi: 10.1016/j.nuclcard.2008.02.009. Epub 2008 Apr 14. PMID 18513639
- [Background] Thomas GS, Tammelin BR, Schiffman GL, Marquez R, Rice DL, Milikien D, Mathur V. Safety of regadenoson, a selective adenosine A2A agonist, in patients with chronic obstructive pulmonary disease: A randomized, double-blind, placebo-controlled trial (RegCOPD trial). J Nucl Cardiol. 2008 May-Jun;15(3):319-28. doi: 10.1016/j.nuclcard.2008.02.013. Epub 2008 Apr 14. PMID 18513638
- [Background] Iskandrian AE, Bateman TM, Belardinelli L, Blackburn B, Cerqueira MD, Hendel RC, Lieu H, Mahmarian JJ, Olmsted A, Underwood SR, Vitola J, Wang W; ADVANCE MPI Investigators. Adenosine versus regadenoson comparative evaluation in myocardial perfusion imaging: results of the ADVANCE phase 3 multicenter international trial. J Nucl Cardiol. 2007 Sep-Oct;14(5):645-58. doi: 10.1016/j.nuclcard.2007.06.114. PMID 17826318
- [Background] Gordi T, Frohna P, Sun HL, Wolff A, Belardinelli L, Lieu H. A population pharmacokinetic/pharmacodynamic analysis of regadenoson, an adenosine A2A-receptor agonist, in healthy male volunteers. Clin Pharmacokinet. 2006;45(12):1201-12. doi: 10.2165/00003088-200645120-00005. PMID 17112296
- [Background] Hendel RC, Bateman TM, Cerqueira MD, Iskandrian AE, Leppo JA, Blackburn B, Mahmarian JJ. Initial clinical experience with regadenoson, a novel selective A2A agonist for pharmacologic stress single-photon emission computed tomography myocardial perfusion imaging. J Am Coll Cardiol. 2005 Dec 6;46(11):2069-75. doi: 10.1016/j.jacc.2005.05.097. Epub 2005 Nov 9. PMID 16325044

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: A: Dobutamine Test Then Regadenoson Test: Arm A will get Dobutamine Stress test with cardiac MR (CMR). Both arms will then cross over to the other arm to get the second test. So each participant will undergo two types of testing.
- Active Comparator: B Regadenoson Test Then Dobutamine: Arm B will get Regadenoson stress test with CMR. Both arms will then cross over to the other arm to get the second test. So each participant will undergo two types of testing.
Period: First Intervention
Arm/Group | Active Comparator: A: Dobutamine Test Then Regadenoson Test | Active Comparator: B Regadenoson Test Then Dobutamine
Started | 10 | 4
Completed | 9 | 3
Not Completed | 1 | 1
Not completed — Did not meeting inclusion/exclusion | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Second Intervention
Arm/Group | Active Comparator: A: Dobutamine Test Then Regadenoson Test | Active Comparator: B Regadenoson Test Then Dobutamine
Started | 9 | 3
Completed | 6 | 3
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Sample: Overall Study Sample
Arm/Group | Overall Study Sample
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 69 [57 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Duration of Procedures
Description: To compare the time involved during pharmacologic stress testing using regadenoson versus intravenous dobutamine in individuals with moderate to severe chronic obstructive pulmonary disease (COPD)or asthma.
Time Frame: 1 day
Measure: Mean (Full Range); unit: Minutes
Groups:
- Dobutamine: All participants that completed Dobutamine testing
- Regadenoson: All participants that completed the regadenoson testing
Arm/Group | Dobutamine | Regadenoson
Number analyzed (Participants) | 12 | 9
Minutes | 48 [35 to 75] | 55 [28 to 138]

2. Secondary Outcome: Ease of Administration of Regadenoson Versus Intravenous Dobutamine Using Compare MD Questionnaire
Description: The Compare MD tool have the following scales: Ease of Administration - Scale from 1(most easy among all MRI stress tests) to 5(most difficult), low score represent better outcome. Patient Comfort - Scale from 1(very comfortable) to 4(very uncomfortable), low score represent better outcome. Interruptions during the procedure - Scale from 1(1-2) to 4(>6), low score represent better outcome. Side effects - Scale from 1(fewer than any other MRI stress test) to 4(the most), low score represent better outcome. Level of anxiety while during the procedure - Scale from 1(less than any other MRI stress test) to 4(the most), low score represent better outcome. Overall rating of the procedure (1 very Difficult to 5 very easy), higher scores represent better outcomes.
Time Frame: 1 day
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Dobutamine | Regadenoson
Number analyzed (Participants) | 12 | 9
units on a scale
  Ease of administration | 2.9 [1 to 4] | 1.9 [1 to 3]
  Patient Comfort | 1.8 [1 to 3] | 1.5 [1 to 3]
  Interruptions during the procedure | 0.5 [0 to 1] | 0.1 [0 to 1]
  Side effects | 2.3 [1 to 3] | 1.6 [1 to 2]
  Level of anxiety while during the procedure | 2.4 [1 to 3] | 1.5 [1 to 3]
  Overall rating of the procedure | 4.3 [2 to 5] | 4.1 [3 to 5]

3. Secondary Outcome: Ease of Administration of Regadenoson Versus Intravenous Dobutamine Using Compare MD Questionnaire (Episodes of Arrhythmias, Bradycardia, and Wheezing)
Description: Ease of Administration of regadenoson versus intravenous dobutamine using Compare MD Questionnaire. Episodes of arrhythmias (including PVCs) and bradycardia (HR<60), low score represent better outcome. Number of Episodes of wheezing and SPO2<94%, low numbers represent better outcome.
Time Frame: 1 day
Measure: Mean (Full Range); unit: number of episodes
Arm/Group | Dobutamine | Regadenoson
Number analyzed (Participants) | 12 | 9
number of episodes
  Episodes of arrhythmias and bradycardia | 0.6 [0 to 4] | 0.1 [0 to 1]
  Episodes of wheezing and SPO2<94% | 0.0 [0 to 0] | 0.0 [0 to 0]

4. Secondary Outcome: Ease of Administration of Regadenoson Versus Intravenous Dobutamine Using Compare Tech Questionnaire
Description: To compare the ease of administration of regadenoson verses intravenous dobutamine during pharmacological stress testing in individuals with moderate to severe chronic obstructive pulmonary disease (COPD) or asthma. Patient Comfort - Scale from 1(very comfortable) to 4(very uncomfortable), low score represent better outcome. Interruptions during the procedure - Scale from 1(1-2) to 4(>6), low score represent better outcome. Level of monitoring - Scale from 1(most easy among all MRI tests) to 4(most difficult), low score represent better outcome. Level of anxiety while during the procedure - Scale from 1(less than any other MRI stress test) to 4(the most), low score represent better outcome. Overall rating of the procedure - Scale from 1(very difficult) to 4(very easy), higher scores represent better outcome.
Time Frame: 1 day
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Dobutamine | Regadenoson
Number analyzed (Participants) | 12 | 9
units on a scale
  Patient Comfort | 1.2 [0 to 3] | 1.5 [1 to 3]
  Interruptions during the procedure | 0.6 [0 to 2] | 0.1 [0 to 1]
  Level of monitoring | 2.7 [1 to 4] | 1.1 [0 to 2]
  Level of anxiety while during the procedure | 1.8 [1 to 3] | 1.3 [0 to 2]
  Overall rating of the procedure | 3.5 [2 to 5] | 4.3 [4 to 5]

5. Secondary Outcome: Ease of Administration of Regadenoson Versus Intravenous Dobutamine Using Compare Tech Questionnaire (Episodes of Wheezing)
Description: To compare the ease of administration of regadenoson verses intravenous dobutamine during pharmacological stress testing in individuals with moderate to severe chronic obstructive pulmonary disease (COPD) or asthma. Low scores represent better outcome.
Time Frame: 1 day
Measure: Mean (Full Range); unit: number of episodes
Arm/Group | Dobutamine | Regadenoson
Number analyzed (Participants) | 12 | 9
number of episodes | .2 [0 to 1] | 0.0 [0 to 0]

6. Secondary Outcome: Ease of Administration of Regadenoson Versus Intravenous Dobutamine Using Compare Nurse Questionnaire
Description: To compare the ease of administration of regadenoson verses intravenous dobutamine during pharmacological stress testing in individuals with moderate to severe chronic obstructive pulmonary disease (COPD) or asthma. Ease of Administration - Scale from 1(most easy among all MRI stress tests) to 5(most difficult), low score represent better outcome. Patient Comfort - Scale from 1(very comfortable) to 4(very uncomfortable), low score represent better outcome. Interruptions during the procedure - Scale from 1(1-2) to 4(>6), low score represent better outcome. Side effects - Scale from 1(fewer than any other MRI stress test) to 4(the most), low score represent better outcome.
Time Frame: 1 day
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Dobutamine | Regadenoson
Number analyzed (Participants) | 12 | 9
units on a scale
  Ease of administration | 3.4 [2 to 5] | 1.5 [1 to 2]
  Patient Comfort | 2.3 [1 to 4] | 1.5 [1 to 2]
  Interruptions during the procedure | 0.6 [0 to 2] | 0.1 [0 to 1]
  Side effects | 2.0 [1 to 3] | 1.3 [1 to 2]

7. Secondary Outcome: Ease of Administration of Regadenoson Versus Intravenous Dobutamine Using Compare Nurse Questionnaire (Episodes of Arrhythmias, Bradycardia, Hypertension, and Wheezing)
Description: To compare the ease of administration of regadenoson verses intravenous dobutamine during pharmacological stress testing in individuals with moderate to severe chronic obstructive pulmonary disease (COPD) or asthma. Episodes of (SBP>140), low number represent better outcome. Episodes of arrhythmias (including PVCs) and bradycardia (HR<60), low number represent better outcome. Episodes of wheezing and SPO2<94%, low number represent better outcome.
Time Frame: 1 day
Measure: Mean (Full Range); unit: number of episodes
Arm/Group | Dobutamine | Regadenoson
Number analyzed (Participants) | 12 | 9
number of episodes
  Episodes of hypertension | 1.6 [0 to 7] | 2 [0 to 8]
  Episodes of arrhythmias and bradycardia | .8 [0 to 4] | .8 [0 to 4]
  Episodes of wheezing and SPO2<94% | 0.0 [0 to 0] | 0.0 [0 to 0]

ADVERSE EVENTS:
Arm/Group | Dobutamine | Regadenoson
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 0/9 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dobutamine (N=9) | Regadenoson (N=3)
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Severe headache that persisted for 2 days.
Abdominal Complaints (Gastrointestinal disorders) | 0 (0) | 1 (1) — Abdominal complaints, reminiscence of reactivation of Irritable Bowel Syndrome. Referred to specialist

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No